CLINICAL TRIAL: NCT06049238
Title: Comparison of Post Facilitation Stretch and Maitland Mobilization in Improving Range of Motion in Post-traumatic Stiff Elbow
Brief Title: Comparison of Post Facilitation Stretch and Maitland Mobilization in Post-traumatic Stiff Elbow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCRAHS-ISB/REC/MS-PT/01608
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Post Traumatic Stiff Elbow
Keywords: Post facilitation stretch.; Maitland.; Stiff elbow

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maitland Mobilization (Experimental): Maitland mobilization will be applied 2-3 oscillations per second for 1 minute, 5 set each day, 5 days a week for 4 weeks.
  Interventions: Other: Maitland Mobilization
- post facilitation stretch (Active Comparator): PFS will be performed 6-10s isometric contraction with 100 % force followed by 15s passive stretch, 4-5 repetitions per day, 5 days a week for 4 weeks.
  Interventions: Other: Post facilitation stretch

INTERVENTIONS:
Other: Maitland Mobilization — * Hot Pack for 10 mints
  * Active and active-assisted exercises (10 reps x 3 sets) for the
  * Elbow flexion and extension
  * Wrist flexion and extension
  * Forearm supination and pronation
  Arms: Maitland Mobilization
Other: Post facilitation stretch — * Hot Pack for 10 mints
  * Active and active-assisted exercises (10 reps x 3 sets) for the
  * Elbow flexion and extension
  * Wrist flexion and extension
  * Forearm supination and pronation
  Arms: post facilitation stretch

SUMMARY:
This research study aims to bridge the gap in the existing literature by comparing the efficacy of Maitland mobilization and PFS techniques in the treatment of post-traumatic stiff elbow. While existing research has shown the favorable effects of joint mobilization and muscle energy techniques in other musculoskeletal conditions, there is a notable gap in understanding their efficacy in post-traumatic stiff elbow, particularly in Pakistan where no such study has been conducted. By investigating the comparative outcomes of these techniques, this research will contribute valuable clinical insights, potentially guiding clinicians in selecting the most effective treatment approach and laying the foundation for evidence-based treatment protocols tailored to patients with post-traumatic stiff elbow.

DETAILED DESCRIPTION:
The elbow being a highly constrained synovial hinge joint has a high propensity for degeneration and stiffness. There could be functional losses seen with even less severe loss of range of motion (ROM) at the elbow. The stiff or contracted elbow is defined as an elbow with a reduction in extension greater than 30 degrees, and/or a flexion less than 120 degrees. Although supination and pronation are often reduced as well, this will not be considered further as contracture of the elbow is not related to forearm rotation. The elbow is more prone to stiffness because Brachialis muscle lies directly over the anterior capsule, the anterior capsule tends to tear more frequently than posterior, all 3 elbow articulations exist in 1 capsule, the elbow is prone to development of Heterotrophic Ossification. Loss of terminal extension is less disabling than loss of the same degree of terminal flexion. It was a randomized, controlled trial, conducted among post-traumatic stiff elbow patients. Sample size was 32 by using G Power Calculator. Participants were randomly assigned to the intervention or control group after a baseline assessment with a lottery ticket and an opaque envelope. All participants in both groups were evaluated on two occasions: (i) baseline (ii) After 4 weeks of intervention

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 35 years
* Both male and female
* Patients with a limitation of elbow joint range of motion greater than 30 degrees in extension and less than 120 degrees in flexion.
* 2-3 months after POP, splinting
* Patients having bone ossification on X-ray findings will be included.

Exclusion Criteria:

* Patients with a history of rheumatoid arthritis or other inflammatory joint diseases
* Mal-union or non- union elbow fracture.
* Patients with a history of neuromuscular disorders or other conditions affecting muscle tone.
* Patients with a history of previous elbow surgery or joint replacement.
* Patients with a history of traumatic brain injury or other neurological conditions affecting upper limb function.
* Patients with open reduction
* Patient with elbow dislocation
* Elbow joint mal-alignment
* Heterotopic ossification
* Myositis ossification or posttraumatic ankyloses.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 4 weeks
  Changes from baseline Numeric pain rating scale is a self-administered, or analyst reported, measuring instrument comprising of a scale that shows numerical ranges usually from 0-10 or 0-100. In this scale extreme or farthest point shows having 'no pain' to having 'extreme pain'.
ROM Elbow (Flexion) | 4 weeks
  Changes from baseline range of motion( ROM) of elbow joint flexion is taken by using Goniometer.
ROM Elbow (Extension) | 4 weeks
  Changes from baseline range of motion( ROM) of elbow joint extension is taken by using Goniometer.
ROM Forearm (Supination) | 4 weeks
  Changes from baseline range of motion( ROM) of forearm supination is taken by using Goniometer.
ROM Forearm (Pronation) | 4 weeks
  Changes from baseline range of motion (ROM) of forearm pronation is taken by using Goniometer.

SECONDARY OUTCOMES:
Disability | 4 weeks
  Changes from baseline disability is measured through DASH (Disability of the arm, shoulder and hand) questionnaire. DASH questionnaire is a self reported area specific outcome measuring tool for symptoms and disabilities in upper limb. It mainly comprise of a 30-items scale which is further consist of questions related to difficulty in performing normal daily activities, scored on 5 response options. Scores for these 30 items then calculate on a scale of 0 (no disability) to 100 (most severe disability)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia ishtiaq, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No